CLINICAL TRIAL: NCT00783861
Title: Study for Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability, Dermical Sensitivity) of Dermacyd Femina Pocket BR.
Brief Title: Dermacyd Femina (Lactic Acid) Pocket BR - Compatibility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04370
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Lactic Acid (Dermacyd Femina)
  Interventions: Drug: Lactic Acid

INTERVENTIONS:
Drug: Lactic Acid — Lactic Acid (Dermacyd Femina)

SUMMARY:
To demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd Femina (Lactic Acid) Pocket BR.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 60 years old;
* Phototype Skin I,II, III e IV
* Integral skin test in the region;
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion;

Exclusion criteria:

* Lactation or gestation
* Use of Antiinflammatory and/or immunosuppression drugs one month before the study;
* Personnel history of atopy;
* History of sensitivity or irritation for topic products;
* Active cutaneous disease;
* Use of new drugs or cosmetics during the study;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The absence of primary and accumulated dermical irritability and dermical sensitivity will be evaluated using International Contact Dermatitis Research Group (ICDRG) scale. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com